CLINICAL TRIAL: NCT04098133
Title: Epidemiology of Carbapenemase-producing Bacteria in a Swiss Tertiary Care Hospital
Acronym: CPB-Epi Basel
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-01548; me19Tschudinsutter
Record Dates: First submitted 2019-09-17; First posted 2019-09-23 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Infections With CPB
Keywords: Carbapenemase-producing Klebsiella pneumoniae; antibiotic resistancy; infections with Carbapenemase-producing Bacteria (CPB); Carbapenemase-producing Bacteria
MeSH Terms: interventions — Data Collection; Demography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: data collection for demographic data — data collection for demographic data (age, gender, hospital admission and discharge date, length of stay, hospitalization prior to current hospital stay (acute care facilities, long-term healthcare centres, nursing homes), discharge destination, outcome, cause of death, travel history, previous exposure to antibiotics and proton pump Inhibitors)
Other: data collection for clinical data — data collection for clinical data (comorbidities, Charlson Comorbidity Index, immunosuppressive treatment, date of diagnosis of CPB, days between hospital admission and diagnosis of CPB, type of consecutive infection, indwelling vascular hardware, urinary catheterization, surgical therapies)
Other: data collection for treatment data — data collection for treatment data (antibiotic therapy, immunosuppressive therapy, concomitant medication)
Other: data collection for microbiological data — data collection for microbiological data (species of CPB, type of sample, date of sample, history of colonization or infection with any antibiotic resistant pathogen)

SUMMARY:
This retrospective and prospective study is to investigate the incidence of Carbapenemase-producing bacteria (CPB) at the University Hospital Basel, the time to detection of CPB and to initiation of infection control measures, the risk factors associated with carriage of CPB, type and duration of previously administrated antibiotic medication, antibiotic treatment, as well as to assess the outcomes of the affected patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with detection of carbapenemase-producing bacteria from January 1st , 2008 until December 31st , 2028

Exclusion Criteria:

* Patients with documented refusal of subsequent use of their data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated in the in- or outpatient setting at the University Hospital Basel with detection of carbapenemase-producing bacteria in any screening or clinical sample from January 1st , 2008 until December 31st , 2028
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-08-22 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
incidence of CPB at the University Hospital Basel (number) | from January 1st , 2008 until December 31st, 2028
  incidence of CPB at the University Hospital Basel (number)

SECONDARY OUTCOMES:
time to detection of CPB (days) | from January 1st , 2008 until December 31st, 2028
  time to detection of CPB (days)
time to initiation of infection control measures | from January 1st , 2008 until December 31st, 2028
  time to initiation of infection control measures
time to adequate treatment in patients with CPB infections | from January 1st , 2008 until December 31st, 2028
  time to adequate treatment in patients with CPB infections
presence of established risk factors for CPB | from January 1st , 2008 until December 31st, 2028
  presence of established risk factors for CPB
length of hospital stay (days) | from January 1st , 2008 until December 31st, 2028
  length of hospital stay (days)
discharge destination | from January 1st , 2008 until December 31st, 2028
  discharge destination
cure from infection | from January 1st , 2008 until December 31st, 2028
  cure from infection
cause-specific mortality (number) | from January 1st , 2008 until December 31st, 2028
  cause-specific mortality (number)
all-cause mortality (number) | from January 1st , 2008 until December 31st, 2028
  all-cause mortality (number)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Tschudin Sutter, Prof. Dr. MD, Principal Investigator — University Hospital Basel, Division of Infectious Diseases and Hospital Epidemiology
Locations (1):
- Division of Infectious Diseases and Hospital Epidemiology, Basel, Switzerland